CLINICAL TRIAL: NCT06495541
Title: The Real World Study of Pyrotinib in the Treatment of Advanced Breast Cancer With HER2 Positive
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tianjin Cancer Hospital..
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; RWS; Pyrotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib (Other)
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Administration method: Pyrrolitinib standard dose: 400 mg once a day, oral administration within 30 minutes after breakfast, continuous administration for 21 days per cycle. The dosage can be determined by the doctor according to the actual situation Make adjustments. Other medications: The doctor selects the medication plan based on the actual situation.

SUMMARY:
Research object：Planned to receive pyrrolidine for HER2 positive first-line breast cancer patients

Research purpose:

Main research objectives:

To observe the efficacy and safety of pyrrolidine in the treatment of HER2 positive advanced first-line breast cancer.

Secondary research objectives:

1. Evaluate the correlation between patient characteristics in the late stage of treatment and specific treatment plans and clinical outcomes Sex (including safety outcomes)
2. Evaluate whether and how previous anti HER2 therapy affects the efficacy of subsequent pyrrolitinib treatment
3. To observe the efficacy of pyrrolitinib in patients with brain metastasis of HER2 positive breast cancer

Research endpoint:

Main research endpoint:

Progression free survival (rwPFS)

Secondary study endpoint:

Efficacy endpoints: objective response rate (rwORR), disease control rate (rwDCR), until treatment failure Time to Flight (TTF), Total Survival (OS), Security

DETAILED DESCRIPTION:
Overall Study Design: This study adopts a prospective, multicenter, and observational design, with a planned enrollment of 500 first-line patients who plan to receive pyrrolitinib treatment for HER2 positive patients. The medication regimen is not restricted, Fully follow the clinical choices of doctors and evaluate the clinical benefits of using different modes of pyrrolitinib (PFS) and security. The imaging evaluation is based on the RECIST 1.1 standard and is conducted by reference to the The research center conducts tumor efficacy evaluation. Patients using pyrrolitinib need to undergo a safety visit on the 28th day of the last administration, and thereafter Enter survival follow-up until patient death or trial termination (whichever occurs first).

Administration method: Pyrrolitinib standard dose: 400 mg once a day, oral administration within 30 minutes after breakfast, continuous administration for 21 days per cycle. The dosage can be determined by the doctor according to the actual situation Make adjustments. Other medications: The doctor selects the medication plan based on the actual situation.

Inclusion criteria:

1. Age ≥ 18 years old;
2. Pathological or histopathological confirmed HER2 positive cases cannot be surgically advanced or metastasized Patients with sexual breast cancer (HER2 positive is defined as: standard immunohistochemistry (IHC) Detected as 3+or ISH positive);
3. There is a traceable medical history record during the treatment period;
4. Voluntarily participate in this study, sign informed consent, have good compliance, and are willing to cooperate Follow up.

Exclusion criteria:

1. Failure to sign informed consent form;
2. Previous history of other malignant tumors, but cured skin basal cell carcinoma and cervical cancer Excluding cancer;
3. Difficulty in swallowing, chronic diarrhea, and intestinal obstruction, which can affect medication administration and absorption Various factors;
4. Pregnant or lactating women, and women of childbearing age who cannot achieve optimal contraception;
5. Any other circumstances in which the researcher deems the patient unsuitable to participate in this study.

Research principle: In the first-line treatment of HER2 positive breast cancer with pyrrolitinib, trastuzumab and docetaxel, the median PFS assessed by the investigator as the primary endpoint was 24.3 months, and the ORR was 88%.

Approved by the National Medical Products Administration (NMPA) for HER2 positive in April 2023 First line treatment of sexual breast cancer and all indications of pyrrolidine will be covered by medical insurance in 2024 Cover. Pyrrolitinib is currently registered for research and development in neoadjuvant, adjuvant, and advanced stages The research is currently underway, all of which are RCT studies, but there is currently no real-world data available I hope to further verify the efficacy of pyrrolitinib in treating HER2 positive advanced first-line breast cancer in the real world The efficacy and safety of adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Pathological or histopathological confirmed HER2 positive cases cannot be surgically advanced or metastasized Patients with sexual breast cancer (HER2 positive is defined as: standard immunohistochemistry (IHC) Detected as 3+or ISH positive);
3. There is a traceable medical history record during the treatment period;
4. Voluntarily participate in this study, sign informed consent, have good compliance, and are willing to cooperate Follow up.

Exclusion Criteria:

1. Failure to sign informed consent form;
2. Previous history of other malignant tumors, but cured skin basal cell carcinoma and cervical cancer Excluding cancer;
3. Difficulty in swallowing, chronic diarrhea, and intestinal obstruction, which can affect medication administration and absorption Various factors;
4. Pregnant or lactating women, and women of childbearing age who cannot achieve optimal contraception;
5. Any other circumstances in which the researcher deems the patient unsuitable to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 24.3months
  The time from randomization to disease progression evaluated by researchers for patients